CLINICAL TRIAL: NCT07314463
Title: The Effect of Laughter Yoga-Based Mental Health Strengthening Training Applied to Mothers With Children With Special Needs on Caregiving Burden, Positive Mental Health, Perceived Stress and Salivary Cortisol Level
Brief Title: The Psychobiological Effects of Laughter Yoga: An Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Özlem Erdem, PhD, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24112002
Record Dates: First submitted 2025-12-06; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Caregiver; Education
Keywords: Laughter Yoga; Strengthening Mental Health; Caregiver Burden; Positive Mental Health; Stress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Strengthening mental health (Experimental): The intervention group was divided into two subgroups, each consisting of ten participants. Based on participants' availability, the first group's sessions were scheduled for Tuesdays and the second group's sessions for Thursdays. The reason for dividing The intervention group was divided because the mothers were only available on specific days. This arrangement aimed to ensure more effective participation in the training process and enhance group interaction for more efficient implementation of the training. The same interaction-based intervention was implemented in both intervention subgroups with identical content and formats.
  Interventions: Behavioral: Laughter Yoga-Based Mental Health Strengthening Training
- No İntervention (No Intervention): Participants in the control group were asked to complete a Personal Information Form, the Zarit Caregiver Burden Scale, the Positive Mental Health Scale, and the Perceived Stress Level Scale. Participants in the control group received no intervention. Cortisol saliva samples were collected from participants in the control group simultaneously with the experimental group. Posttests were taken from participants in the control group after the intervention sessions.

INTERVENTIONS:
Behavioral: Laughter Yoga-Based Mental Health Strengthening Training — This laughter yoga-based training program is distinct from traditional practices because of its structured psychoeducational content. In addition to laughter exercises, it aims to enhance participants' self-awareness, stress management, and communication skills through informative and reflective sessions. Each session began with cognitive and emotional awareness-building activities, followed by physical laughter practices, promoting mind-body integration. Thus, the program offers multidimensional benefits, including emotional relief, cognitive development, social skill enhancement, and strengthening internal coping resources.
  Arms: Experimental: Strengthening mental health

SUMMARY:
This study was conducted to determine the effect of Laughter Yoga-Based Mental Health Enhancement Training, applied to mothers of children with special needs, on the burden of care, positive mental health, perceived stress, and salivary cortisol levels.

DETAILED DESCRIPTION:
Individuals with special needs are those with physical, developmental, or behavioral differences and require more intensive and specialized care in areas such as education, healthcare, and social life. Mothers, as the primary caregivers of children, play a significant role in meeting the needs of children with special needs. However, the extraordinary effort exerted by these mothers can become challenging due to various circumstances, leading to increased caregiving burden and difficulties in the physical, emotional, social, or economic areas. During this process, mothers may become vulnerable to mental health problems and may need support to cope with these challenges. Therefore, providing empowerment training to protect and improve the mental health of mothers of children with special needs is essential in the future.

This study was a randomized controlled trial designed with a pre-test post-test experimental design. The study group consisted of mothers of children with special needs who were receiving special education at a Rehabilitation Center in Konya, Turkey. A total of 40 participants were included in the study: 20 in the intervention group and 20 in the control group.

Data collection tools included the Personal Information Form, the Zarit Caregiver Burden Scale, the Positive Mental Health Scale, and the Perceived Stress Scale. Saliva samples were also collected to measure the cortisol levels of the participants. The intervention group received an 8-week Laughter Yoga-Based Mental Health Empowerment Training, administered by the researcher. No intervention was provided to the control group (CG).

Before the study began, ethical approval was obtained from the Non-Invasive Clinical Research Ethics Committee of a university's Faculty of Nursing, institutional permission was received from the Provincial Directorate of National Education, and written informed consent was obtained from all participants.

For data analysis:

* Independent Sample t-tests were used to compare numerical descriptive variables between groups,
* Pearson's chi-square and Fisher's exact tests were used for categorical variables.
* Pearson's correlation coefficients were used to examine the relationships between numerical variables.
* Mixed-design ANOVA was used to compare changes over time within the groups.
* Logistic regression analysis was conducted to determine the significant predictors in the intervention group.
* The strength of the relationship between the dependent and independent variables in the logistic regression was evaluated using Cox-Snell R² and Nagelkerke R².
* A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being the primary caregiver of the child
* Having a score of 21 or higher on the Zarit Caregiver Burden Scale
* Understanding and speaking Turkish at a level sufficient to complete data collection forms and participate in sessions

Exclusion Criteria:

* Having participated in a similar program within the last 6 months

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women were chosen as biological mothers
Enrollment: 40 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Zarit Caregiving Burden Scale | 8 weeks after the initial assessment
  It is used to assess the emotional, social, and physical burden an individual experiences as a result of their caregiver role.
Positive Mental Health Scale | 8 weeks after the initial assessment
  It is used to define and assess positive mental health.
Perceived Stress Scale | 8 weeks after the initial assessment
  It is used to determine the extent to which individuals perceive certain events in their lives as stressful.
Salivary cortisol levels | Every week for 8 weeks
  There will be a relationship between laughter yoga-based mental health strengthening training and mothers' salivary cortisol levels.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu K UYAROĞLU, Associate Professor, Study Director — Selcuk University; Özlem ERDEM, MSC, Principal Investigator — Selcuk University
Locations (1):
- Directorate of National Education, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided